CLINICAL TRIAL: NCT05333705
Title: Trial of Donor Immune Cell Therapy for Acute Myeloid Leukemia.
Brief Title: Donor Immune Cell Therapy for Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJYFY-2020N8
Record Dates: First submitted 2022-03-23; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2021-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: natural killler cell; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Study Arms: Experimental arm: Cytokine Arm Infusions of Natural Killer (NK) cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- immune cell arm (Experimental): Umbilical cord blood or donated peripheral blood of healthy donors were collected and NK cells were cultured. NK cell production will be infused after chemotherapy.
  Interventions: Biological: infusion of natural killer cells

INTERVENTIONS:
Biological: infusion of natural killer cells — Umbilical cord blood or donated peripheral blood of healthy donors were collected and NK cells were sorted and cultured. NK cell production will be infused after chemotherapy

SUMMARY:
This study aims to introduce a new technology of donor NK cell infusion. NK cells defend against viruses and cancer cells in vivo whereas this effect declines in patiens with tumors. In this study, NK cells will be separated from donated peripheral blood or umbilical cord blood. Eligible NK cells will be infused to patients with Acute myeloid leukemia (AML). This new therapy will probably induce their sustained remission and reduce recurrences.

DETAILED DESCRIPTION:
Primary end point:

To determine the rate of overall survival at 2 years of Interventional cohort

Secondary end point:

To determine the cumulative incidence of relapse at 2 years. To determine the rate of disease-free survival at 2 years. Describe the safety and toxicity of donor NK cell infusion.

Study Design:

This study is a phase I clinical trial. 15 eligible AML patients will be enrolled sequentially to receive detached NK cells product during induction or consolidation therapy. Refractory or relapsed patients and patients who achieved complete remission (CR) after induction therapy are included. They will receive anthracycline-based chemotherapy according to NCCN guidelines. At the same time, Cultured NK cells will be infused into patients after chemotherapy. Anti-allergic therapy and prophylaxis of graft versus host disease (GVHD) will be given before infusion. Treatment effect will be measured and adverse effect will be treated and documented after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been diagnosed as acute myeloid leukemia in accordance with "Chinese Diagnosis and Treatment Guidelines of AML". Those who achieved CR after chemotherapy are mainly included. Refractory/relapsed AML can also be enrolled.
* Patients with normal heart function (ejection fraction ≥ 50%), normal liver function(ALT and AST ≤ 2.5 times the upper limit of normal value, bilirubin ≤ 2 times the upper limit of normal value) and normal renal function with blood creatinine ≤ 3.0 mg/dL (≤ 260 µmol /L) can be enrolled.
* Patients will be required to sign an informed consent.

Exclusion Criteria:

* Patients with severe infection or other malignant tumors.
* Women during pregnancy or lactation.
* Other patients deemed unsuitable by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
hematological response rate | up to 2 years, from treatment begining to death
  Hematological Complete Remission (HCR): Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0x10^9/L; platelet count >100x10^9/L.
Overall survival | Up to 2 years after beginning treatment
  Overall survival (OS) is measured from the date of first infusion of NK cells to the date of death from any cause; patients not known to have died at last follow up are censored on the date they were last known to be alive.

SECONDARY OUTCOMES:
Cumulative incidence of relapse | Up to 2 years after beginning treatment
  Relapse was defined as the recurrence of above 5%bone marrow blasts and the reappearance of blasts in the blood or the development of extramedullary disease infiltrates at any site.
Disease free survival (DFS) | Up to 2 years after beginning treatment
  Disease free survival (DFS) is defined as the time from the date of first infusion of NK cells to the date of relapse or death as a result of any cause.
Incidence of adverse effects | Up to 2 years after beginning treatment
  Toxic effects were graded according to the National Cancer Institute's Common Toxicity Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: huaiyu Wang, doctor, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruggeri L, Capanni M, Casucci M, Volpi I, Tosti A, Perruccio K, Urbani E, Negrin RS, Martelli MF, Velardi A. Role of natural killer cell alloreactivity in HLA-mismatched hematopoietic stem cell transplantation. Blood. 1999 Jul 1;94(1):333-9. PMID 10381530
- [Background] Miller JS, Soignier Y, Panoskaltsis-Mortari A, McNearney SA, Yun GH, Fautsch SK, McKenna D, Le C, Defor TE, Burns LJ, Orchard PJ, Blazar BR, Wagner JE, Slungaard A, Weisdorf DJ, Okazaki IJ, McGlave PB. Successful adoptive transfer and in vivo expansion of human haploidentical NK cells in patients with cancer. Blood. 2005 Apr 15;105(8):3051-7. doi: 10.1182/blood-2004-07-2974. Epub 2005 Jan 4. PMID 15632206
- [Background] Bachanova V, Cooley S, Defor TE, Verneris MR, Zhang B, McKenna DH, Curtsinger J, Panoskaltsis-Mortari A, Lewis D, Hippen K, McGlave P, Weisdorf DJ, Blazar BR, Miller JS. Clearance of acute myeloid leukemia by haploidentical natural killer cells is improved using IL-2 diphtheria toxin fusion protein. Blood. 2014 Jun 19;123(25):3855-63. doi: 10.1182/blood-2013-10-532531. Epub 2014 Apr 9. PMID 24719405
- [Background] Curti A, Ruggeri L, Parisi S, Bontadini A, Dan E, Motta MR, Rizzi S, Trabanelli S, Ocadlikova D, Lecciso M, Giudice V, Fruet F, Urbani E, Papayannidis C, Martinelli G, Bandini G, Bonifazi F, Lewis RE, Cavo M, Velardi A, Lemoli RM. Larger Size of Donor Alloreactive NK Cell Repertoire Correlates with Better Response to NK Cell Immunotherapy in Elderly Acute Myeloid Leukemia Patients. Clin Cancer Res. 2016 Apr 15;22(8):1914-21. doi: 10.1158/1078-0432.CCR-15-1604. Epub 2016 Jan 19. PMID 26787753